CLINICAL TRIAL: NCT03780985
Title: Hang-up Versus Non-fixation Technique for Immediate Post-placental Intrauterine Device Insertion During Cesarean Section
Brief Title: Post-placental Intrauterine Device Insertion During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mahmoud Mohammed, Assistant Lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUD-Zahraa
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Intrauterine Device Migration
MeSH Terms: conditions — Intrauterine Device Migration | interventions — Cesarean Section; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrauterine device insertion with a suture fixation (Active Comparator): Intruterine device through hysterotomy incision during cesarean section with a suture fixation
  Interventions: Procedure: Intrauterine device insertion; Procedure: Cesarean section; Procedure: Suture
- intrauterine device insertion without a suture fixation (Active Comparator): IUD through hysterotomy incision during cesarean section without a suture fixation
  Interventions: Procedure: Intrauterine device insertion; Procedure: Cesarean section

INTERVENTIONS:
Procedure: Intrauterine device insertion — Post-placental insertion of intrauterine device during Cesarean section
Procedure: Cesarean section — to delivery of the fetus
Procedure: Suture — to fix the intrauterine device
  Arms: intrauterine device insertion with a suture fixation

SUMMARY:
Effective, reversible postpartum contraception decreases the chance of rapid repeat pregnancy and poor perinatal outcome in a subsequent pregnancy especially in women delivered by cesarean section.The traditional 6-week postpartum visits not evidenced based and may not meet patient needs, particularly with respect to provision of contraception.Intrauterine device placement after delivery of the placenta is an appealing strategy for increasing access to postpartum Intrauterine device because it does not require a separate postpartum visit.

Advantage of post-placental Intrauterine device insertion, Intrauterine devices are recommended as first-line contraceptives by the American Academy of Pediatricians. The Centers for Disease Control and Prevention united state . Medical Eligibility Criteria for Contraceptive Use places no restrictions on use, and states advantages generally outweigh the risks for immediate postpartum use of Intrauterine devices.

ELIGIBILITY:
Inclusion Criteria:

1. Age group : 18-40 years
2. Women who will be willing to undergo elective cesarean section
3. women desire using Copper IUD as long acting contraceptive method.

Exclusion Criteria:

1. Intrauterine infection.
2. Fundal Myoma.
3. Hemorrhagic disorder
4. Genital tract malignancy
5. Uterine atony
6. Sexually transmitted infection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of displaced intrauterine device after insertion in both groups | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided